CLINICAL TRIAL: NCT01165021
Title: An Exploratory Phase 2 Study of Pemetrexed/Cisplatin as Pre-operative Chemotherapy in the Treatment of Stage IIIAN2 Nonsquamous Non-Small Cell Lung Cancer
Brief Title: A Study of Pemetrexed/Cisplatin as Pre-operative Treatment of Early Stage Nonsquamous Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13621; H3E-EW-JMIP (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-07-14; First posted 2010-07-19 (Estimated); Results first posted 2014-05-21 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Cisplatin; Folic Acid; Vitamin B 12; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pemetrexed + Cisplatin (Experimental)
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Folic Acid; Drug: Vitamin B12; Drug: Dexamethasone

INTERVENTIONS:
Drug: Pemetrexed — 500 milligram per square meter (mg/m²) administered as an intravenous infusion on Day 1 of 21-day cycles, for 3 cycles
  Other Names: Alimta; LY231514
Drug: Cisplatin — 75 mg/m² administered as an intravenous infusion on Day 1 of 21-day cycles, for 3 cycles
Drug: Folic Acid — Administered orally.
Drug: Vitamin B12 — Administered Intramuscular injection.
Drug: Dexamethasone — Administered orally.

SUMMARY:
The purpose of this trial is to assess how well the combination of pemetrexed with cisplatin can reduce tumor size.

ELIGIBILITY:
Inclusion Criteria:

* Nonsquamous Non-Small Cell Lung Cancer that was confirmed by tissue biopsy
* Stage IIIAN2 disease (T1aN2, T1bN2, T2aN2, T2bN2, and T3N2)
* Tumor considered potentially resectable
* Good performance status (score of 0 or 1) according to Eastern Cooperative Oncology Group scale (ECOG)
* No prior therapy for lung cancer
* Measurable disease according to version 1.1 of Response Evaluation Criteria in Solid Tumors (RECIST) Criteria
* Life expectancy of at least 6 months
* Organs are functioning well (bone marrow reserve, liver, kidney, lung)
* Signed Informed Consent
* Women must be surgically sterile, postmenopausal, or compliant with a medically approved contraceptive regimen (for example, intrauterine device, birth control pills, or barrier device) during and for 6 months after last dose of study drug; must have a negative pregnancy test within 7 days before study enrollment; and must not be breast-feeding.
* Men must be surgically sterile, or compliant with a contraceptive regimen during and for 6 months after last dose of study drug.
* Be fit for surgery at the time of enrollment

Exclusion Criteria:

* Receiving or have received an investigational drug or device within the last 30 days
* Have previously completed or withdrawn from this study or any other study investigating pemetrexed
* Serious concomitant systemic disorder
* Serious cardiac condition, such as myocardial infarction within 6 months, angina, or heart disease
* Receiving concurrent administration of any other anticancer therapy
* Have received a recent (within 30 days of enrollment) or are receiving concurrent yellow fever vaccination
* Inability or unwillingness to take Pemetrexed supplementation/premedication (folic acid, vitamin B12, or corticosteroids)
* Inability to interrupt aspirin or other nonsteroidal anti-inflammatory agents, other than an aspirin dose less than or equal to 1.3 grams per day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-11; Primary Completion 2013-07 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- Italy (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Novara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orbassano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Padua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pisa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sondalo

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant Flow reports participants who discontinued from study treatment. Completed participants were those who had a baseline tumor assessment, finished 3 cycles (Cy) of pre-operative chemotherapy (chemo), and had a second tumor assessment following chemo.
Groups:
- Pemetrexed + Cisplatin: Pemetrexed: 500 milligrams per square meter (mg/m²) administered as an intravenous infusion on Day 1 of 21-day cycles, for 3 cycles
  Cisplatin: 75 mg/m² administered as an intravenous infusion on Day 1 of 21-day cycles, for 3 cycles
Period: Overall Study
Arm/Group | Pemetrexed + Cisplatin
Started | 19
≥1 Dose Chemo | 19
≥1 Dose Chemo, Baseline, Cy 3 Assessment | 17
3 Cycles of Chemo, Then Surgery | 15
Completed | 18
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of chemotherapy.
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (9.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 13
Race/Ethnicity, Customized [Number; unit: participants]
  White | 19
Region of Enrollment [Number; unit: participants]
  Italy | 19
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — ECOG classifies participants according to their functional impairment. Scores range from 0 (fully active) to 5 (death). 0 (fully active, able to carry on all pre-disease performance without restriction) and 1 (restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature).
  participants
    0 | 15
    1 | 4
Initial Pathological Diagnosis [Number; unit: participants] — Initial cancer diagnosis confirmed by tissue biopsy.
  participants
    Adenocarcinoma, Lung | 17
    Carcinoma, Large Cell, Lung | 1
    Carcinoma, Non-Small Cell, Lung | 1
Tumor-Node-Metastasis (TNM) Stage of Disease [Number; unit: participants] — Tumor size: T1=surrounded by lung or visceral pleura with no evidence of invasion more proximal than lobar bronchus; T1a ≤2 centimeters (cm) at greatest dimension (GD); T1b >2 cm, ≤3 cm at GD; T2=involves main bronchus, ≥2 cm distal to carina; invades visceral pleura, associated with atelectasis or obstructive pneumonitis extends to hilar but not entire lung; T2a >3 cm, ≤5 cm at GD; T2b >5 cm, ≤7 cm at GD; T3= >7 cm or 1 that invades the thoracic cavity. Nodal status (N): N2 =Metastasis in ipsilateral mediastinal and/or subcarinal lymph nodes. Distant metastasis (M): M0 =No distant metastasis.
  participants
    T1aN2M0 | 3
    T1bN2M0 | 2
    T2aN2M0 | 3
    T2bN2M0 | 3
    T3N2M0 | 8
Tobacco Consumption Status [Number; unit: participants]
  Current Tobacco User | 4
  Former Tobacco User | 12
  Never Used Tobacco | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) [Overall Response Rate (ORR)]
Description: Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST v1.1) criteria. CR was defined as the disappearance of all target and non-target lesions and all target and non-target lymph nodes were non-pathological or normal in size [<10 millimeter (mm) short axis]. PR was defined as having at least a 30% decrease in sum of longest diameter of target lesions taking as reference the baseline sum diameters. ORR calculated as: (sum of the number of participants with PRs and CRs) divided by (number of evaluable participants) multiplied by 100.
Time Frame: From study enrollment until disease progression or recurrence up to completion of 3 cycles (21-day cycles) of chemotherapy
Population: Participants who received at least 1 dose of preoperative chemotherapy and had baseline and Cycle 3 scans for tumor assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 17
percentage of participants | 41.2 [18.4 to 67.1]

2. Secondary Outcome: Percentage of Participants With No Viable Tumor Cells in Resected Lung Tissue [Pathological Complete Remission (pCR)]
Description: pCR after the participant has undergone surgery was calculated as: (total number of participants with pCR) divided by (the total number of participants in pathological response population) multiplied by 100.
Time Frame: At the time of surgery (within 3 to 6 weeks of Day 1 of Cycle 3 [21-day cycles] of chemotherapy)
Population: Participants who received at least 1 dose of preoperative chemotherapy and had surgical tumor tissue samples available.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 15
percentage of participants | 93.3 [68.1 to 99.8]

3. Secondary Outcome: Percentage of Participants Who Exhibit a Downward Shift in Tumor Extent From Stage IIIAN2 to Stages IIIA, II, I, or Stage 0
Description: Tumor downstaging compared to baseline (Stage IIIAN2) were those participants who exhibited a downward shift in tumor extent from Stage IIIAN2 to Stages IIIA, II, I, or 0 were reported. Downstaging was based on radiological examination. Stage IIIAN2 was locally advanced and/or involved lymph nodes, metastasis in ipsilateral mediastinal and or subcarinal lymph nodes, tumors were ≤2 centimeters (cm) up to 5 cm in greatest dimension; Stage IIIA was locally advanced and/or involved lymph nodes, tumor extension was restricted to the affected lung; Stage II was locally advanced and/or involved lymph nodes; Stage I was small localized cancers, usually curable; Stage 0 the cancer did not spread beyond the inner lining of the lung. Missing responses were also reported. Percentage of participants calculated as: (number of participants with a downward shift in extent of their tumor) divided by (total number of evaluable participants) multiplied by 100.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 17
percentage of participants
  No Change or Worsening of Tumor Stage | 29.4 [10.3 to 56.0]
  Change to Stage IIIA | 29.4 [10.3 to 56.0]
  Change to Stage II | 11.8 [1.5 to 36.4]
  Change to Stage I | 17.6 [3.8 to 43.4]
  Missing | 11.8 [1.5 to 36.4]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as duration from the date of study enrollment to the date of death from any cause. Participants not known to have died as of the data inclusion cut-off date were censored at the date of last contact. The last contact for participants in post-discontinuation was the last date participant was known to be alive.
Time Frame: Enrollment until the date of death from any cause up to 64 months
Population: All participants who received 1 or more doses of preoperative chemotherapy. Participants censored=8
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 19
months | 34.6 [10.8 to NA] — Upper range of 95% confidence interval were not calculated due to high censoring rate.

5. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from date of first dose to the first observation of disease progression or death due to any cause. For participants not known to have died or did not have objective progressive disease (PD) as of the data inclusion cut-off date, PFS was censored at the date of the last objective progression-free disease assessment. PD was defined using RECIST v1.1 criteria as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (including the baseline sum if that is the smallest). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: Enrollment until the first date of objectively determined PD or death up to 64 months
Population: All participants who received 1 or more doses of preoperative chemotherapy. Participants censored=3.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 19
months | 12.4 [7.0 to 21.7]

ADVERSE EVENTS:
Arm/Group | Pemetrexed + Cisplatin
Serious Adverse Events (participants affected / at risk) | 2/19
Other Adverse Events (participants affected / at risk) | 15/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed + Cisplatin (N=19)
Acute abdomen (Gastrointestinal disorders) | 1 (1)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed + Cisplatin (N=19)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Apical granuloma (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (5)
Oral dysaesthesia (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 3 (3)
Fatigue (General disorders) | 4 (7)
Irritability (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 3 (3)
Bronchitis (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (6)
Platelet count decreased (Investigations) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Depressive symptom (Psychiatric disorders) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cafe au lait spots (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
Due to difficulties identifying suitable participants and enrollment delays, entries were closed after 26 of planned 33 participants signed consent. Results based on 19 participants who received ≥1 dose of chemotherapy. View results with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days